CLINICAL TRIAL: NCT03696667
Title: Affect Regulation Based on Brain-computer Interface Towards Treatment for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mental Health, Singapore (Other)
Collaborators: Agency for Science, Technology and Research (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017/00297
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-09

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affective BCI training (Active Comparator): 15 participants in the intervention group will undergo 24 sessions of BCI-based emotion regulation training over an 8-week period. Each session will take about 30-minute to complete where participants will listen to music with audio feedback to regulate emotions toward positive affect.
  Interventions: Device: BCI
- Control group (No Intervention): 15 participants in the control group will take part in 24 music sessions (with no audio feedback) over an 8-week period. Each session will take about 30-minute to complete.

INTERVENTIONS:
Device: BCI — As participants listen to the music, the EEG waves of their affective states and their variations detected in real-time is converted into an auditory signal providing direct feedback to participants about their affective states and assisting participants to learn and practice emotion regulation.
  Arms: Affective BCI training

SUMMARY:
The primary objective is to examine the feasibility and efficacy of a locally developed brain-computer interface (BCI) based system training for regulating mood in healthy elderly. The investigators hypothesize that elderly who complete the training program will be better at regulating emotions as compared to controls, based on their ratings of the primary outcome measures.

DETAILED DESCRIPTION:
In this project, we will leverage on a locally developed electroencephalograph (EEG)-based BCI technology for decoding affective states of the brain, and thereby develop a closed-loop sensing and stimulation mechanism. The technology uses advanced neural signal computing on the EEG in real-time and audio feedback using a machine learning model that associates individual user's EEG characteristics in relation to music-emotion features. The system is portable and will allow emotion regulation training to be done outside of hospital setting with ease thus potentially addressing the treatment gap for MDD in the elderly.

This is a two group randomized study. One group will undergo the intervention which is 24 sessions of BCI emotion regulation training (i.e. listening to music with audio feedback to regulate emotions towards positive affect) over an 8-week period. The control group will undergo 8 weeks of music sessions, without any emotion regulation training. Both groups will undergo pre- and post- psychometric assessments looking at cognition, quality of life, functioning and emotional states. This study will also carry out functional MRI of the brain before and after 8 weeks of either training (intervention) or music music session (control) to examine changes associated with the affective BCI training. Study findings derived from psychometric assessments, EEG analysis and neuroimaging will provide evidences on efficacy and usability of this technology.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Geriatric Depression Scale score of 4 and below
* Fit to provide informed consent
* Able to travel to study site independently

Exclusion Criteria:

* Presence of hearing impairment
* Presence of any known neuropsychiatric disorders (e.g. dementia, epilepsy or mental retardation)
* Contraindications for MRI such as surgical clips, cardiac pacemakers, metal implants and plates, orthodontics and claustrophobia

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Emotion regulation questionnaire (ERQ) | Week 0 and Week 9
  To evaluate change in ERQ scores
Positive and Negative Affect Scale (PANAS) | Week 0 and Week 9
  To evaluate change in PANAS score

SECONDARY OUTCOMES:
Brief Assessment of Cognition - Short form | Week 0 and Week 9
  To evaluate changes in neurocognition
Geriatric Depression Scale (GDS) | Week 0 and Week 9
  To evaluate change in GDS score
Positive Mental Health (PMH) instrument | Week 0 and Week 9
  To evaluate change in PMH score
Body Awareness Questionnaire (BAQ) | Week 0 and Week 9
  To evaluate change in BAQ
Subjective Happiness Scale | Week 0 and Week 9
  To evaluate change in SHS
Connor-Davidson Resilience Scale 25 (CD-RISC-25) | Week 0 and Week 9
  To evaluate change in CD-RISC-25 score
The Frenchay Activities Index (FAI) | Week 0 and Week 9
  To evaluate change in FAI scores
Medical Outcomes Study: 20-item short form survey instrument | Week 0 and Week 9
Outcome rating scale | After each BCI session during Weeks 1 to 8
Usability questionnaire | At the end of Week 8
  Participants in the intervention group will rate statements regarding their satisfaction and ease of use of the training components on a 7-point Likert scale

OTHER OUTCOMES:
Changes in functional MRI | Week 0 and Week 9
  To examine the neural mechanism underlying the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Lee, Principal Investigator — Institute of Mental Health, Singapore
Locations (2):
- Singapore (2):
  - Duke-NUS Medical School, Singapore
  - Institute of Mental Health, Singapore

IPD SHARING:
Plan to Share IPD: No